CLINICAL TRIAL: NCT04034979
Title: Evaluation of a Context-adapted Decision Aid Supporting Critically Ill Patients' Decisions About Life-sustaining Therapies - a Pilot Project
Brief Title: Evaluation of a Decision Aid About Life-sustaining Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Patrick Archambault, Assistant professor, Laval University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Catalyst-2017-001
Record Dates: First submitted 2018-02-24; First posted 2019-07-29 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Decision Making; Resuscitation; Intensive Care Unit; Goals-of-care; Shared-decision Making
Keywords: decision aid; ICU; goals-of-care; videotaping; shared-decision making
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: 4 phases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I-Baseline evaluation (No Intervention): The first two months of the investigator's project will be a baseline evaluation of the current decision making process about goals-of-care in a local ICU setting (Levis, Quebec). A PhD student will collect sociodemographic data (age, gender, education level, religion), observe and video record (or audio record) dyads of physicians and newly admitted elderly patients discussing goals-of-care.
- Phase II-Impact of the decision aid (Experimental): The two following months will be an evaluation of the decision making process about goals-of-care in the same local ICU setting using only the decision aid without any training. A PhD student will collect sociodemographic data (age, gender, education level, religion), observe and video record (or audio record) new dyads of physicians and newly admitted elderly patients discussing goals-of-care, whether the physician chooses to use the context-adapted decision-aid or not.
  Interventions: Behavioral: decision aid
- Phase III- Impact of the decision aid and the (Experimental): This phase will be an evaluation of the decision making process about goals-of-care in the same local ICU setting after intensivists complete the training program and using the DA. A PhD student will collect sociodemographic data (age, gender, education level, religion), observe and video record (or audio record) new dyads of physicians and newly admitted elderly patients discussing goals-of-care using the context-adapted decision aid and the new skills learned in the training program.
  Interventions: Behavioral: decision aid

INTERVENTIONS:
Behavioral: decision aid — One hour online training about shared-decision making about goals-of-care and best practices regarding goals-of-care discussions and decision-making. One hour debriefing in presence.
  Other Names: training session
  Arms: Phase II-Impact of the decision aid; Phase III- Impact of the decision aid and the

SUMMARY:
Introduction: Clinical practice guidelines recommend shared decision making (SDM) to facilitate goals-of-care discussions. This study will train clinicians about how to use a context-adapted decision aid (DA) and SDM to conduct goals-of-care discussions with the elderly. The objectives of this study are to: 1) determine if the use of the DA and SDM training program: a) increase clinicians' engagement of patients in decision making regarding their goals of care; b) increase adoption of evidence-based behaviours regarding goals-of-care decision making; and 2) identify patients' most frequent incomprehension, concerns, questions and clinicians' opportunities to improve the skills in goals-of-care decision making.

Methods: This study will have three phases. Phase I (May-June 2017) will be a baseline evaluation of the current goals-of-care decision making process with elderly patients in a single ICU setting (Levis, Quebec). Phase II (July-August 2017) will be an evaluation of the goals-of-care decision making process in the same ICU using a DA. Phase III (September-December 2017) will be the delivery of an online and in-person training session about the use of the DA and about how to conduct discussions about goals-of-care. The study will then evaluate the goals-of-care decision making process after completion of the training program and using the DA. The investigators will observe and audio- or video-record all eligible elderly-intensivist dyads discussing goals of care during each phase. Two investigators will analyse the recordings using the OPTION 12 scale (measuring the extent that clinicians engage patients in SDM) and the ACCEPT quality indicators (measuring the extent to which intensivists engage in best practice goals-of-care discussions). The investigators will conduct qualitative content analysis of the video and audio records to identify patients' most frequent incomprehension, concerns, questions and clinicians' opportunities to improve the goals-of-care decision-making skills.

Deliverables: This study will produce evidence regarding the impact of a context-adapted DA and training program on clinicians' adoption of SDM and other best practice behaviors regarding goals-of-care decision making with the elderly, and evidence regarding the most frequent patients' incomprehension, concerns, questions and clinicians' opportunities to improve the goals-of-care decision-making skills.

ELIGIBILITY:
Inclusion Criteria:

1. aged 65 and older,
2. capable of making their own healthcare decisions as determined by the attending intensivist's clinical judgment,
3. in need of a discussion about goals of care as determined by the attending intensivist's clinical judgment.

Exclusion Criteria:

1. intubated patients,
2. patients facing urgent decisions,
3. patients cared by the principal investigator,
4. patients who do not read or speak French.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Observing Patient Involvement in Decision Making (OPTION) scale | The OPTION scale will be measured at the earliest possible time during the patients' intensive care stay (eg., first 24 hours after admission or whenever the patient is capable of engaging in a goals-of-care discussion).
  The OPTION scale (12 items) measures the extent that clinicians engage patients in shared decision making. For each item, a score 0 (The behaviour is not observed) to 4 (The behaviour is observed and executed to a high standard) is given. Adding each item's score will arrive at a number between 0 (minimum) and 48 (maximum). The OPTION scale will be measured by two observers rating audio- or video-recordings of goals-of-care discussions conducted by intensivists with their patients at the earliest possible time during the patients intensive care stay. These discussions will be held at the discretion of the attending intensivist when deemed appropriate. Most often these discussions are held at the time of patient admission (first 24 hours) or whenever the patient is capable of engaging in a goals of care discussion (eg., after the patient is extubated and weaned off mechanical ventilation).
Score based on the quality indicators from the Audit of Communication, Care Planning, and Documentation (ACCEPT) study | The quality indicators will be measured at the earliest possible time during the patients' intensive care stay (eg., first 24 hours after admission or whenever the patient is capable of engaging in a goals-of-care discussion.
  This measure will be based on 7 of the 34 (ACCEPT) quality indicators that measure the quality of end-of-life communication and decision making: written information provided before discussion about goals of care, poor prognosis shared with patient during the discussion, verification with patient about prior discussions or written documents about the use of life-sustaining treatments, use of information by intensivist about about goals of care to support the decision, verification by the intensivist prior to the discussion of any written advanced directives in the patient's medical record, documentation of the goals of care discussed in medical record after discussion, goals of care documented in the medical chart after discussion consistent with patient's stated preferences. Indicators will be measured by two observers rating audio- or video-recordings. Score is the sum of the quality indicator items divided by the sum of highest possible values of these items on a scale 0% to 100%.

SECONDARY OUTCOMES:
Qualitative content analysis | The audio and video recordings will be done at the earliest possible time during the patients' intensive care stay (eg., first 24 hours after admission or whenever the patient is capable of engaging in a goals-of-care discussion.
  Each audio or video recording will be content analysed by a doctoral student and a research assistant using the R language Qualitative Data Analysis (RQDA) package for Qualitative Data Analysis. The aim of this content analysis will be to identify: 1) patients' most frequent incomprehension, concerns, questions and 2) clinicians' opportunities to improve their skills in goals-of-care discussions and decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Archambault, MD, MSc., Principal Investigator — Laval University
Locations (1):
- Centre de recherche de l'Hôtel-Dieu de Lévis, Lévis, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinuff T, Dodek P, You JJ, Barwich D, Tayler C, Downar J, Hartwick M, Frank C, Stelfox HT, Heyland DK. Improving End-of-Life Communication and Decision Making: The Development of a Conceptual Framework and Quality Indicators. J Pain Symptom Manage. 2015 Jun;49(6):1070-80. doi: 10.1016/j.jpainsymman.2014.12.007. Epub 2015 Jan 24. PMID 25623923
- [Background] Heyland DK, Barwich D, Pichora D, Dodek P, Lamontagne F, You JJ, Tayler C, Porterfield P, Sinuff T, Simon J; ACCEPT (Advance Care Planning Evaluation in Elderly Patients) Study Team; Canadian Researchers at the End of Life Network (CARENET). Failure to engage hospitalized elderly patients and their families in advance care planning. JAMA Intern Med. 2013 May 13;173(9):778-87. doi: 10.1001/jamainternmed.2013.180. PMID 23545563
- [Background] Heyland D, Cook D, Bagshaw SM, Garland A, Stelfox HT, Mehta S, Dodek P, Kutsogiannis J, Burns K, Muscedere J, Turgeon AF, Fowler R, Jiang X, Day AG; Canadian Critical Care Trials Group; Canadian Researchers at the End of Life Network. The Very Elderly Admitted to ICU: A Quality Finish? Crit Care Med. 2015 Jul;43(7):1352-60. doi: 10.1097/CCM.0000000000001024. PMID 25901550
- [Background] Kon AA, Davidson JE, Morrison W, Danis M, White DB; American College of Critical Care Medicine; American Thoracic Society. Shared Decision Making in ICUs: An American College of Critical Care Medicine and American Thoracic Society Policy Statement. Crit Care Med. 2016 Jan;44(1):188-201. doi: 10.1097/CCM.0000000000001396. PMID 26509317
- [Background] Legare F, Stacey D, Turcotte S, Cossi MJ, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for improving the adoption of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2014 Sep 15;(9):CD006732. doi: 10.1002/14651858.CD006732.pub3. PMID 25222632
- [Background] Evans R, Edwards A, Brett J, Bradburn M, Watson E, Austoker J, Elwyn G. Reduction in uptake of PSA tests following decision aids: systematic review of current aids and their evaluations. Patient Educ Couns. 2005 Jul;58(1):13-26. doi: 10.1016/j.pec.2004.06.009. PMID 15950832
- [Background] White DB, Braddock CH 3rd, Bereknyei S, Curtis JR. Toward shared decision making at the end of life in intensive care units: opportunities for improvement. Arch Intern Med. 2007 Mar 12;167(5):461-7. doi: 10.1001/archinte.167.5.461. PMID 17353493
- [Derived] Plaisance A, Turgeon J, Souza LG, Legare F, Turcotte S, Germain N, Jean T, Dionne M, Fortier FA, Plante P, Tapp D, Gelinas V, Belanger E, Ebell MH, Chabot C, van de Belt TH, Turgeon AF, Archambault PM. Exploring the Impact of a Context-Adapted Decision Aid and Online Training About Shared Decision Making About Goals of Care with Elderly Patients in the Intensive Care Unit: A Mixed-Methods Study. Patient. 2026 Jan;19(1):145-160. doi: 10.1007/s40271-025-00761-7. Epub 2025 Sep 25. PMID 40999300